CLINICAL TRIAL: NCT04022551
Title: Emergency Room Evaluation and Recommendations for Older Users of Emergency Departments: a Cohort Study Database on the Effects of ER2 Recommendations on Length of Stay and Hospital Admission
Brief Title: Emergency Room Evaluation and Recommendations for Older Users of Emergency Departments
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1851
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Elderly Care; Length of Hospital Stay; Multimorbidity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: At Emergency nurses will carry out a test called: Emergency Room Evaluation and Recommendation which contents the following statements:
  1. Being 85 years older and over (Yes/No)
  2. Male (Yes/No)
  3. Home services (Yes/No)
  4. Taking 5 different medication daily (Yes/No)
  5. Use of walking aid (Yes/No)
  6. Disoriented (Yes/No)

SUMMARY:
The study evaluates if the Emergency Room Evaluation and Recommendation Tool (ER2) reduces the hospital admission rate and the length of stay in Emergency.

DETAILED DESCRIPTION:
Regardless of the reason for ED visit and its care plan, there are simple interventions, which may be continued to prevent short-term ED adverse outcomes. Delirium, motor deconditioning, adverse drug reactions due to polypharmacy, and inappropriate home support are the main conditions to target when taking care of older ER users.

Evidence based medicine showed that simple and early intervention in the process of care may prevent delirium (e.g., hydration, avoid restraint, mobilize and satisfy basic needs, time and place reorientation) and motor deconditioning (e.g., encourage mobility, up to chair at meal time during day light hours, provide appropriate walking aid) in older patients. The medication reconciliation is also an efficient intervention for the prevention of adverse drug reactions. Furthermore, an early assessment of home support is a crucial step to adjust home services for an early discharge to home.

ELIGIBILITY:
Inclusion Criteria:

* Being 75 years old and over
* Being brought at Emergency on medical stretcher

Exclusion Criteria:

* Being less than 75 years old
* Never come at Emergency

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: It will be enrolled participants who are 75 years and over, and who will be brought at Emergency on medical stretcher. At Emergency, nurses will carry out a test called: Emergency Room Evaluation and Recommendation.
Sampling Method: Non-Probability Sample
Enrollment: 4724 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospital admission rate by age | Around 10 months
  The recommendation of the Emergency Room Evaluation Tool will be used to reduce the hospital admission rate in older at Emergency.

SECONDARY OUTCOMES:
Length of stay at Emergency | Around 10 months
  The recommendation of the Emergency Room Evaluation Tool will be used to reduce the length of stay at Emergency.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada